CLINICAL TRIAL: NCT00580021
Title: Clinical Outcomes in Hereditary Cancer
Status: Withdrawn | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-004
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer; Pancreatic Cancer
Keywords: Ashkenazi ancestry; mutations in BRCA1 or BRCA2; Breast Cancer; Pancreatic Cancer
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Once potential subjects are identified, pathology records will be reviewed to establish which of the potential subjects have archived pathology material available at MSKCC. It is important to note that the material does not have to be tumor and, in fact, benign tissue, such as uninvolved lymph node, will be sought by preference. However, tumor tissue will be used if no benign tissue is available.

GROUPS / COHORTS (1):
- 1: Patients with breast and pancreas cancer.
  Interventions: Other: Genotyping

INTERVENTIONS:
Other: Genotyping — Samples for DNA extraction will be shaved from archival paraffin-embedded tissue blocks (using normal lymph node preferentially)and placed in appropriate receptacles labeled only with the subject unique study number. This material will be transported to the genotyping laboratory, where it will be stored until the clinical record abstraction is complete. Briefly, DNA will be extracted from the archive paraffin-embedded material using standard protocols and the samples will be analyzed for the presence of the Ashkenazi BRCA founder mutations using either PCR-based or gel-electrophoresis-based approaches.

SUMMARY:
Compare the clinical characteristics and post-surgical outcomes (overall survival)of pancreatic cancer patients of Ashkenazi descent with or without germline founder mutations in BRCA1 or BRCA2 .

Compare the clinical characteristics and outcomes (time to progression) of breast cancer patients of Ashkenazi descent with or without germline founder mutations in BRCA1 or BRCA2 receiving paclitaxel chemotherapy for metastatic disease.

DETAILED DESCRIPTION:
Compare the clinical characteristics and post-surgical outcomes (overall survival)of pancreatic cancer patients of Ashkenazi descent with or without germline founder mutations in BRCA1 or BRCA2 .

Compare the clinical characteristics and outcomes (time to progression) of breast cancer patients of Ashkenazi descent with or without germline founder mutations in BRCA1 or BRCA2 receiving paclitaxel chemotherapy for metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Included in DB0363-03
* Jewish religious preference at registration
* Archival material available for testing
* Adequate post-surgical follow-up
* Jewish religious preference at registration
* Archival material available for testing
* Adequate follow-up to determine time to progression

Exclusion Criteria:

-Subjects will not be included in the analyses if a DNA sample cannot be obtained.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects will be individuals with the disease of interest during the time period of interest who described their religious preference at the time of registration to be Jewish.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The overall objective of the protocol is to examine the hypothesis that hereditary cancers are distinct in clinical characteristics and outcome from those that arise in the absence of a known predisposition. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org